# Comparison of Patient Satisfaction Between Conventional and Digital Removable Partial Dentures

# NCT Number NCT0722898828

APRIL 15, 2025

**Patient Consent** 

# KINGDOM OF SAUDI ARABIA Ministry Of Education

### KING ABDULAZIZ UNIVERSITY

FACULTY OF DENTISTRY University Dental Hospital



# المملكة العربية السعودية ورزارة التعليم المعة الملك عود العزيز كلية طب الأسنان مستشفى الأسنان الجامعي

# إقرار بالموافقة على المشاركة في الدراسة

# عنوان الدراسة: النتائج المتعلقة بالمرضى للأطقم الجزئية المصنوعة من معدن الكروم كوبالت المصبوب أو ثلاثي الأبعاد المطبوع أو من مادة البولي ايثر ايثر كيتون. تجربة سريرية عشوائية

| معلومات الطبيب المعالج | معلومات المريض |
|---|---|
| اسم الطبيب المعالج: | اسم المريض: |
| القسم: لاستعاضة السنية | رقم الملف الطبي: |
| 18 17 16 15 14 13 12 11 Appell Condition of the state of | 21 22 23 24 25 26 27 28 Augil Left Upper 1 2 3 4 5 6 7 8 Left Lover 4 4 5 6 7 8 Left Lover 4 4 5 6 7 8 Left Lover 4 4 5 6 7 8 Left Lover 4 5 6 7 8 Left Lover |

في حال موافقتك على الانضمام لهذه الدراسة فسوف نقوم بعمل ثلاثة أنواع مختلفة من الأطقم الجزئية المتحركة المصنوعة من مواد و طرق مختلفة و ذلك لقياس مدى رضا المريض عن كل نوع و تأثير هذه الأطقم على جودة الحياة المتعلقة بصحة الفم و الأسنان . سوف تستعمل كل نوع من هذه التركيبات لمدة شهر ثم تمتنع عن استعمال اي منها لمدة اسبوع كنوع من الراحة مما يساعدك على اعادة تقييم النوع التالي. في نهاية كل مرحلة من العلاج اي بعد شهر من استعمال التركيبة ستقوم بتعبئة استبيان يتضمن مجموعة من الاسنلة تقيم مدى رضاك عن التركيبة خلال فترة الاستعمال و مدى تأثيرها على الحياة المتعلقة بصحة الفم و الأسنان.

#### المضاعفات و المخاطر

لايوجد أي مضاعفات أو مخاطر حقيقية او جوهرية مترتبة على استعمال أيا من انواع الأطقم المتحركة الثلاثة المستعملة في هذه الدراسة. فقط قد تشعر بعدم الارتياح او التوائم مع التركيبة في بداية الاستعمال و هذا سيقل تدريجيا مع الوقت، اذا شعرت بأي ألم من المشابك أو عدم تطابق العضة بشكل كامل فيمكنك اخبار الطبيب لتحسين وضع التركيبة حتى تختفي هذه المشاكل

#### القه ائد٠

ستحصل نتيجة الانضمام لهذه الدراسة على ثلاثة أطقم متحركة مختلفة كلها مصنوعة بحرفية تامة و بدون أي مقابل مادي. هذه الدراسة ستساعد في اختيار الاطقم المتحركة الاكثر مناسبة و ارضاءا للمريض.

#### السرية:

جميع معلوماتك و بياناتك و اجاباتك على الاستبيانات ستكون في سرية تامة و لن يطلع عليها أحد. سيعطى لك رقم يدون على جميع الاوراق الخاصة بك دون ظهور اسمك عليها.

# الانسحاب من الدراسة:

في حال قررت الانسحاب من للدراسة في أي وقت يمكنك ذلك براحة تامة و بدون أي شروط أو تأثير على علاجك بالمستشفى

## التواصل مع الباحث:

في حال كان لديك أي أسئلة يمكنك التواصل مع الباحث الرئيسي لاي استفسار او اذا واجهت أي مشكلة عن طريق الايميل التالي: emesallum@kau.edu.sa

| | ••••• | • | | | افر انا |
|---|---|---|---|---|---|
| على هذا أوقع | ، الانضمام لها و | انني او افق علم | ة بهذه الدر اسة و | المعلومات الخاصا | انني قر أت |

توقيع المريض: \_\_\_\_\_\_ التاريخ: \_\_\_\_\_

#### KING ABDULAZIZ UNIVERSITY

FACULTY OF DENTISTRY University Dental Hospital







### **Informed Consent Form (English Version)**

Study Title: Patient related outcomes of conventional cast Cr-CO, 3D printed Cr-Co, and PEEK removable partial dentures. A randomized clinical trial

#### **Procedures**

If you agree to participate in this study, three removable partial dentures will be made for you, each using a different material (cast Co–Cr, 3D-printed Co–Cr, and PEEK). You will use each denture for 30 days. Between each denture, there will be a one-week rest period. At the end of each period, you will be asked to answer two questionnaires about your satisfaction and oral health related factors.

#### **Potential Risks**

There are no expected serious risks associated with this study. Some participants may experience temporary mild discomfort or adaptation difficulties when wearing a new denture. If any irritation or discomfort occurs, adjustments will be provided immediately.

#### **Benefits**

There will be no financial compensation for participation. However, you will receive three professionally fabricated removable partial dentures free of charge. The results of this study may help improve the quality of removable denture treatment in the future.

## **Confidentiality**

All information collected in this study will be kept strictly confidential. Your name will not appear in any reports or publications. Each participant will be identified only by a study number.

## **Voluntary Withdrawal**

Your participation in this study is completely voluntary. You have the right to refuse to participate or to withdraw at any time without giving a reason. Your decision will not affect your future dental care or relationship with the Faculty of Dentistry.

#### **Contacts for Questions**

If you have any questions or concerns about the study, you may contact the Principal Investigator using the following Email: emesallum@kau.edu.sa

#### **Consent Statement**

| I have read and understood the information above. | I voluntarily agree to participate in this study. |
|---|---|

| Participant's Name: | |
|---------------------|-------|
| Signature: | Date: |
| _ | |